CLINICAL TRIAL: NCT04199065
Title: Impact of the Implementation of Good Practice Guidelines on Beliefs-attitudes and Behavior in the Face of Evidence-based Practice and on the Perception of the Nurses' Work Environment
Brief Title: Impact of Good Practice Guidelines on Evidence-based Practice and Nurses' Work Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); COIB, Col·legi d'Infermers i infermeres de Barcelona (Unknown); Department of Health, Generalitat de Catalunya (PERIS) (Unknown)
Responsible Party: Principal Investigator, Silvia Esteban, RN, MsC, PhD, Parc de Salut Mar
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEIm-PSMAR 2018/8087/I
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Nurses' Work Environment; Committed Centers With Excellence in Care (CCEC®) Program; Nurses' Evidence-based-practice Attitudes; Nurse Physician Relations; Practice Nurse's Scope; Professional Stress
Keywords: Evidence-Based Practice; nurses' Workplace; Good Practices Guides; Hospital
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good Practice Guidelines group (Experimental): Implementation of Good Practice Guidelines
  Interventions: Other: Good Practice Guidelines implementation
- usual practices group (No Intervention): Not Implementation of Good Practice Guidelines, so working as the usual way

INTERVENTIONS:
Other: Good Practice Guidelines implementation — Implementation of Good Practice Guidelines on the framework of the Best Practice Spotlight Organization in Spain (CCEC® / BPSO®), that allows a standardized methodology for providing care and registering indicators.
  Arms: Good Practice Guidelines group

SUMMARY:
Evidence-based practice (EBP) has improved patient health outcomes. The work environment of nurses is a key element to improving the quality of care and to facilitate EBP, while also improving health outcomes.

The CCEC® / BPSO® program consists of the implementation of Good Practice Guides in health organizations in the Spanish territory, and is carried out through a training and participatory methodology, actively involving nurses in the process.

The present study tries to know if in the health organizations where the CCEC® / BPSO® program has been implemented, the perception of the nurses' working environment has improved, as well as their attitude towards evidence-based practice, with respect to organizations where this program has not been implemented.

DETAILED DESCRIPTION:
Quasi-experimental pre-post multicentre study with a non-equivalent control group, within the framework of the third cohort of the RNAO Good Practice Guidelines Implementation Program in Centers Committed to Care Excellence (CCEC® / BPSO®).

PARTICIPATING INSTITUTIONS:

Intervention group(IG): (institutions included in the third cohort of CCEC®):

Estructura de Gestión Integrada de Lugo, Cervo y Monforte de Lemos (Galicia), Hospital General Universitario Santa Lucía (Murcia), Xerencia de Xestión Integrada de A Coruña (Galicia), Hospital Guadarrama (Madrid), Hospital Universitari Germans Trias i Pujol (Cataluña), Hospital Regional Universitario de Málaga (Andalucía), Organización Sanitaria Integrada OSI Araba (Araba).

Control group(CG): Hospital Son Espases (Mallorca), Hospital Son Llàtzer (Mallorca), Hospital de Granollers (Barcelona), Hospital de Puigcerdà (Girona), Hospital d'Igualada (Barcelona), Hospital General Universitario de Alicante (Alicante), Hospital Comarcal de Vinaròs de Castellón de la Plana (Castellón), Hospital Clínic de Barcelona (Barcelona), Hospital Universitario de Fuenlabrada (Madrid), Hospital de la Santa Creu i Sant Pau (Barcelona).

To collect data, two validated questionnaires will be passed to all nurses in 7 health institutions where the RNAO Good Practice Guidelines Implementation Program begins (experimental group) and in 10 where it is not implemented (control group), both groups distributed throughout the Spanish territory. Basal data will be recorded before the beginning of the program and post intervention data will be recorded after one year.

Then the results will be compared to determine whether there are differences between nurses who work in the group of hospitals that have started the program with respect to those who work in other centers. The total duration of the project will be three years.

ELIGIBILITY:
Inclusion Criteria:

Nurses Work in the institutions participating in the study Acceptance to participate in the study

Exclusion Criteria:

Not be active

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
change in Nurses' work environment | baseline and 1 year
  self reported perceived current work environment through the Practice Environment Scale-Nursing Work Index (PES-NWI) questionaire, with 31 Likert type questions (1: "Strongly Disagree" -> 4 "Strongly Agree"), including 5 sub-scales: Nurse participation in hospital affairs (8 questions); nursing foundations for quality of care (10 questions); nurse manager ability, leadership and support of nurses (5 questions); staffing and resource adequacy (4 questions); and collegial nurse-physician relationships (3 questions)
change in Beliefs- attitudes and behavior in front of EBP | baseline and 1 year
  self-reported Beliefs- attitudes and behavior in front of EBP, through the 60 Likert type questions (from 1: minimum agreement to 10: maximum agreement) of the Health Sciences-Evidence Based Practice questionnaire (HS-EBP), that are classified in 5 dimensions: Beliefs and attitudes, (12 items); Results from scientific research (14 items); Development of professional practice (10 items); Evaluation of results (12 items) and Barriers / Facilitators (12 items).

SECONDARY OUTCOMES:
change in Job satisfaction: Likert type question rating | baseline and 1 year
  self-reported job satisfaction through a unique Likert type question rating 1: very unsatisfied; 5: very satisfied.
change in Institutional attitude perceived by nurses in relation to nursing research | baseline and 1 year
  self-reported 4 question rating: yes, not, unknown.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Esteban-Sepúlveda, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute), Barcelona
Locations (17):
- Spain (17):
  - Organización Sanitaria Integrada (OSI) Araba, Vitoria-Gasteiz, Araba
  - Hospital Universitri Germans Tries i Pujol, Badalona, Barcelona
  - Hospital de Granollers, Granollers, Barcelona
  - Consorci Sanitari Anoia-Hospital Igualada, Igualada, Barcelona
  - Hospital Comarcal de Vinaròs, Vinaròs, Castelló
  - Hospital de Puigcerdà, Puigcerdà, Girona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital de Guadarrama, Guadarrama, Madrid
  - Xerencia de Xestión Integrada de A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clínic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Lucus Augusti, Lugo
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital General Universitario Santa Lucía, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: No
Not considered, since the data processing will be done on an aggregate basis.

REFERENCES:
- [Result] Aiken LH, Sermeus W, Van den Heede K, Sloane DM, Busse R, McKee M, Bruyneel L, Rafferty AM, Griffiths P, Moreno-Casbas MT, Tishelman C, Scott A, Brzostek T, Kinnunen J, Schwendimann R, Heinen M, Zikos D, Sjetne IS, Smith HL, Kutney-Lee A. Patient safety, satisfaction, and quality of hospital care: cross sectional surveys of nurses and patients in 12 countries in Europe and the United States. BMJ. 2012 Mar 20;344:e1717. doi: 10.1136/bmj.e1717. PMID 22434089
- [Result] Aiken LH, Sloane DM, Clarke S, Poghosyan L, Cho E, You L, Finlayson M, Kanai-Pak M, Aungsuroch Y. Importance of work environments on hospital outcomes in nine countries. Int J Qual Health Care. 2011 Aug;23(4):357-64. doi: 10.1093/intqhc/mzr022. Epub 2011 May 11. PMID 21561979
- [Result] Cho E, Chin DL, Kim S, Hong O. The Relationships of Nurse Staffing Level and Work Environment With Patient Adverse Events. J Nurs Scholarsh. 2016 Jan;48(1):74-82. doi: 10.1111/jnu.12183. Epub 2015 Dec 7. PMID 26642177
- [Result] Fernandez-Dominguez JC, de Pedro-Gomez JE, Morales-Asencio JM, Bennasar-Veny M, Sastre-Fullana P, Sese-Abad A. Health Sciences-Evidence Based Practice questionnaire (HS-EBP) for measuring transprofessional evidence-based practice: Creation, development and psychometric validation. PLoS One. 2017 May 9;12(5):e0177172. doi: 10.1371/journal.pone.0177172. eCollection 2017. PMID 28486533
- [Result] Fuentelsaz-Gallego C, Moreno-Casbas MT, Gonzalez-Maria E. Validation of the Spanish version of the questionnaire Practice Environment Scale of the Nursing Work Index. Int J Nurs Stud. 2013 Feb;50(2):274-80. doi: 10.1016/j.ijnurstu.2012.08.001. Epub 2012 Sep 1. PMID 22944284
- [Result] Heater BS, Becker AM, Olson RK. Nursing interventions and patient outcomes: a meta-analysis of studies. Nurs Res. 1988 Sep-Oct;37(5):303-7. PMID 3047692